CLINICAL TRIAL: NCT02793557
Title: A Randomised, Double-blind, Placebo-controlled Trial of FOL-005 to Investigate Clinical Safety and Effect on Hair Growth in Healthy Volunteers
Brief Title: Investigation of FOL-005 on Clinical Safety and Effect on Hair Growth
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Follicum AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FCS-001
Record Dates: First submitted 2016-05-16; First posted 2016-06-08 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Hypertrichosis; Alopecia; Hirsutism
MeSH Terms: conditions — Hypertrichosis; Alopecia; Hirsutism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Intradermal injection of 50 μl solution. One application in SAD part for each dosing occasion. 2 or 3 times weekly for 3 month in MD part.
  Interventions: Other: Placebo
- FOL-005: Solution 1 (Experimental): Intradermal injection of 50 μl solution. One application in SAD part. 2 or 3 times weekly for 3 month in MD part.
  Interventions: Drug: FOL-005
- FOL-005: Solution 2 (Experimental): Intradermal injection of 50 μl solution. One application in SAD part. 2 or 3 times weekly for 3 month in MD part.
  Interventions: Drug: FOL-005
- FOL-005: Solution 3 (Experimental): Intradermal injection of 50 μl solution. One application in SAD part. 2 or 3 times weekly for 3 month in MD part.
  Interventions: Drug: FOL-005
- FOL-005: Solution 4 (Experimental): Intradermal injection of 50 μl solution. One application in SAD part. 2 or 3 times weekly for 3 month in MD part.
  Interventions: Drug: FOL-005

INTERVENTIONS:
Drug: FOL-005 — Intradermal injection of 50 μl solution
  Arms: FOL-005: Solution 1; FOL-005: Solution 2; FOL-005: Solution 3; FOL-005: Solution 4
Other: Placebo
  Arms: Placebo

SUMMARY:
A study to investigate clinical safety and effect on hair growth of FOL-005 in healthy volunteers. The study is divided in two parts, a single ascending dose (SAD) part and a multiple dose (MD) part.

DETAILED DESCRIPTION:
SAD part:

A total of 3 weeks dosing, the two lowest concentrations in week 1, dose 3 at week 2 and finally dose 4 at week 3.

MD part:

In total 12 weeks of dosing where group A will be dosed twice weekly and group B three times weekly

Each injection will be administered into one of five of the six randomized areas (10 cm apart, left and right side) from the subject's defined investigational skin areas. One area will be completely untreated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, aged 18-45 years
* Clinically visible terminal hair growth on thighs

Exclusion Criteria:

* Damaged skin in or around test sites
* History of any acute (e.g. acute infections) or chronic illness or known skin cancer that might confound the results of the trial
* History or clinical signs of keloids or hypertrophic scars
* Immunological disorders such as alopecia areata, and systemic lupus erythematosus
* Current or within 2 weeks prior to first dosing use of vasodilating drugs (e.g. Pentoxifyllin, nitroglycerine) or anticoagulating drugs (e.g. heparine, cumarines, new oral anticoagulants)
* Current or within 3 months prior to first dosing use of anti-inflammatory medication, corticosteroids or immunosuppressive drugs taken for more than 2 consecutive weeks
* Current or within 3 months prior to first dosing use of medication with hair growth modifying properties like minoxidil, diazoxid, cyclosporine, antiandrogens
* Current or within 12 months prior to first dosing intake of anabolics or 5-alpha reductase inhibitors
* Current or within one week prior to first dosing use of any topical drugs on the legs

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability by assessing the number and severity of adverse events after intradermal applications of FOL-005 in healthy subjects | 3 months

SECONDARY OUTCOMES:
Effect of FOL-005, as compared to placebo, with respect to number of hairs/cm2 | 3 months
Effect of FOL-005, as compared to placebo, with respect to proportion of telogen hairs | 3 months
Effect of FOL-005, as compared to placebo, with respect to proportion of anagen hairs | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Blume-Peytavi, Professor, Principal Investigator — Klinik für Dermatologie, Venerologie und Allergologie, Charité-Universitätsmedizin Berlin Charitéplatz 1 - 10117 Berlin
Locations (1):
- Klinik für Dermatologie, Venerologie und Allergologie, Charité-Universitätsmedizin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided